CLINICAL TRIAL: NCT02864368
Title: Peptide Targets for Glioblastoma Against Novel Cytomegalovirus Antigens
Acronym: PERFORMANCE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Eric Thompson, M.D. (Other)
Collaborators: Annias Immunotherapeutics, Inc. (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Eric Thompson, M.D., Assistant Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00034208_1; 2R42CA153845-02 (NIH)
Record Dates: First submitted 2016-07-26; First posted 2016-08-12 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
Keywords: PERFORMANCE; Pro00034208; Cytomegalovirus; Ashley
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 5-day TMZ: Components A and B (Experimental): All patients receive Tetanus-Diphtheria booster vaccine at time of enrollment. Cycles of standard TMZ (150-200 mg/m^2/day on days 1-5 of each 28 day cycle) with PEP-CMV vaccination on Day 23 (-1 day, + 2 days) of each TMZ cycle and tetanus pre-conditioning the day before the first vaccine.
  Interventions: Drug: 5-day TMZ; Biological: PEP-CMV: Component A; Drug: Tetanus-Diphtheria booster; Drug: Tetanus Pre-Conditioning; Biological: PEP-CMV: Component B
- 21-day TMZ: Components A and B (Experimental): All patients receive Tetanus-Diphtheria booster vaccine at time of enrollment. Cycles of dose-intensified TMZ (75-100 mg/m^2/day on days 1-21 of each 28 day cycle) with PEP-CMV vaccination on day 23 (-1 day, + 2 days) of each TMZ cycle and tetanus pre-conditioning the day before the first vaccine.
  Interventions: Drug: 21-day TMZ; Biological: PEP-CMV: Component A; Drug: Tetanus-Diphtheria booster; Drug: Tetanus Pre-Conditioning; Biological: PEP-CMV: Component B
- 5-day TMZ: Safety Cohort (Experimental): All patients receive Tetanus-Diphtheria booster vaccine at time of enrollment. Cycles of standard TMZ (150-200 mg/m^2/day on days 1-5 of each 28 day cycle) with PEP-CMV vaccination on Day 23 (-1 day, + 2 days) of each TMZ cycle and tetanus pre-conditioning the day before the first vaccine. Vaccine components A and B were administered separately, with a delay between them, to determine if it was an individual component or a combination of the components that resulted in adverse reactions.
  Interventions: Drug: 5-day TMZ; Biological: PEP-CMV: Component A; Drug: Tetanus-Diphtheria booster; Drug: Tetanus Pre-Conditioning; Biological: PEP-CMV: Component B
- 5-day TMZ: Component A Alone (Experimental): All patients receive Tetanus-Diphtheria booster vaccine at time of enrollment. Cycles of standard TMZ (150-200 mg/m^2/day on days 1-5 of each 28 day cycle) with PEP-CMV vaccination on Day 23 (-1 day, + 2 days) of each TMZ cycle and tetanus pre-conditioning the day before the first vaccine.
  Interventions: Drug: 5-day TMZ; Biological: PEP-CMV: Component A; Drug: Tetanus-Diphtheria booster; Drug: Tetanus Pre-Conditioning
- 21-day TMZ: Component A Alone (Experimental): All patients receive Tetanus-Diphtheria booster vaccine at time of enrollment. Cycles of dose-intensified TMZ (75-100 mg/m^2/day on days 1-21 of each 28 day cycle) with PEP-CMV vaccination on day 23 (-1 day, + 2 days) of each TMZ cycle and tetanus pre-conditioning the day before the first vaccine.
  Interventions: Drug: 21-day TMZ; Biological: PEP-CMV: Component A; Drug: Tetanus-Diphtheria booster; Drug: Tetanus Pre-Conditioning

INTERVENTIONS:
Drug: 5-day TMZ — Chemotherapy agent FDA approved to treat newly-diagnosed glioblastoma given as cycles of 150-200 mg/m^2/day on days 1-5 of each 28 day cycle
  Other Names: temozolomide; Temodar
  Arms: 5-day TMZ: Component A Alone; 5-day TMZ: Components A and B; 5-day TMZ: Safety Cohort
Drug: 21-day TMZ — Chemotherapy agent FDA approved to treat newly-diagnosed glioblastoma given as cycles of dose-intensified TMZ (75-100 mg/m2/day on days 1-21 of each 28 day cycle)
  Other Names: temozolomide; Temodar
  Arms: 21-day TMZ: Component A Alone; 21-day TMZ: Components A and B
Biological: PEP-CMV: Component A — 500 µg of PEP-CMV Component A (a synthetic long peptide) mixed with Montanide ISA-51 intradermally administered
Drug: Tetanus-Diphtheria booster — At time of enrollment, after signing consent and undergoing immune monitoring blood work, patients will receive Tetanus-diphtheria booster vaccination with 0.5 mL of Td (tetanus, diphtheria toxoid, absorbed)
  Other Names: Td; tetanus
Drug: Tetanus Pre-Conditioning — All patients will receive a tetanus pre-conditioning injection in the right groin intradermally on day 22 (±1 day) of the first post-radiation cycle of TMZ
  Other Names: Td; Tetanus-Diphtheria; tetanus
Biological: PEP-CMV: Component B — 500 µg of PEP-CMV Component B (a neutralizing antibody epitope from human CMV glycoprotein B conjugated to Keyhole Limpet Hemocyanin) mixed in 150 µg of GM-CSF intradermally administered
  Arms: 21-day TMZ: Components A and B; 5-day TMZ: Components A and B; 5-day TMZ: Safety Cohort

SUMMARY:
Newly diagnosed glioblastoma (GBM) patients with complete or partial surgical resection who were CMV seropositive patients were eligible to enroll on this trial. Patients were enrolled following standard of care chemoradiation and prior to initiation of post-radiation cycles of temozolomide (TMZ) provided they met all eligibility criteria. All eligible patients received a tetanus-diphtheria (Td) vaccination. Patients enrolled on study were randomized to receive either standard TMZ or dose-intensified TMZ (excluding the safety cohort who only received standard TMZ). All patients received a pre-conditioning injection of tetanus on day 22 of the first post-radiation cycle of TMZ. The following day, patients received the first of 3 intradermal (i.d.) injections of the study drug cytomegalovirus peptide (PEP-CMV), which contained either a combination of Component A and Component B or Component A only depending upon when they enrolled on study. Vaccines #2 and #3 will be given at 2 week intervals. Patients who were O[6]-methylguanine-DNA methyltransferase (MGMT) unmethylated received one adjuvant cycle of the TMZ regimen according to their assigned TMZ arm. Patients who were MGMT methylated or whose methylation status was inconclusive continue with up to 12 cycles of TMZ. After the completion of a patient's last TMZ cycle, vaccines continued every 4-6 weeks for a maximum number of 20 vaccines (unless tumor progression occurred). The study ended prematurely due to lack of funds. The preliminary results suggest that the vaccine may be capable of generating an immune response.

DETAILED DESCRIPTION:
Patients were enrolled following radiation therapy and prior to initiation of post-radiation therapy cycles of adjuvant TMZ provided they met all eligibility criteria. After signing main consent, patients had immune monitoring blood work collected and received a Tetanus-diphtheria booster vaccination with 0.5 mL of Td (tetanus, diphtheria toxoid, adsorbed). After meeting all eligibility criteria, patients were randomized to receive either standard TMZ (150-200 mg/m^2/day on days 1-5 of each 28-day cycle) with vaccination on Day 23 (-1 day, + 2 days) of each TMZ cycle or to receive dose-intensified TMZ (75-100 mg/m^2/day on days 1-21 of each 28-day cycle) with vaccination on day 23 (-1 day, +2 days) of each TMZ cycle (excluding patients enrolled in the safety cohort who only received standard TMZ).

Patients began their initial cycle of adjuvant TMZ as soon as possible following randomization, if applicable. For Arm 1, the adjuvant TMZ cycle(s) will be given as described above. If a patient had an MGMT unmethylated tumor, they discontinued TMZ after the 1st cycle.

All patients received a tetanus pre-conditioning injection in the right groin on day 22 (+1 day) of cycle 1 of adjuvant TMZ. On the following day, patients receive their study vaccine (either a combination of Component A and Component B or Component A only depending upon when they enrolled on study).

Vaccines #2 and #3 were given at 2 week intervals (+ 3 days), which will resulted in a ~35-day delay before starting TMZ cycle 2. MGMT unmethylated patients did not receive subsequent cycles of TMZ, but continued to receive vaccines approximately every 4 (+2) weeks. Originally, patients received the vaccine as follows: 500 µg of PEP-CMV Component A mixed with Montanide Incomplete Freund's Adjuvant (ISA)-51 intradermally administered in the right groin and 2 hours later, 500 µg of PEP-CMV Component B mixed in 150 µg of Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) intradermally administered in the left groin. A safety cohort was added in 2017 following hypersensitivity reactions in which patient received different schedules of vaccine Components A and B to determine the source of the hypersensitivity reactions. Following this safety cohort, the randomized study was allowed to reinitiate with changes to vaccine administration procedure.

Subsequent revisions were made to the study in the latter part of 2018, due to a continuation of hypersensitivity reactions, and Component B was removed from the study. Patients then received the vaccine as follows: 500 µg of PEP-CMV Component A mixed with Montanide ISA-51 administered intradermally with half in the right groin and half in the left groin.

Patients were imaged with contrast-enhanced magnetic resonance imaging (MRI) within 2 weeks (+3 days) after vaccine 3 and then approximately every 8 weeks. RANO criteria was used for assessment of pseudo-progression, and patients demonstrating definitive progression were removed from study. Blood for immune monitoring was obtained at several time points.

The study ended prematurely due to lack of funds.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histopathologically proven newly-diagnosed primary glioblastoma with complete or partial surgical resection. Biopsy not acceptable.
3. Patients must be cytomegalovirus (CMV) seropositive.
4. The tumor must be supratentorial.
5. Karnofsky performance status of ≥ 70.
6. Stable or decreasing steroid dose (≤ 4 mg/day) at time of post-radiation treatment (XRT) adjuvant TMZ initiation. If patients are decreasing steroid use, once they are at 2 mg/day, they may be supplemented with physiologic replacement hydrocortisone therapy (20-30 mg/day in divided doses), at the discretion of the treating oncologist.
7. Hematology: absolute neutrophil count (ANC) ≥ 1500 cells/µL, Platelet count ≥ 100,000 cells/µL, Hemoglobin ≥ 9.0 g/dl
8. Chemistry: ALT/AST ≤ 3.0 times the upper limit of normal (ULN), Total bilirubin ≤ 1.5 mg x ULN (Exception: Patient has known Gilbert's Syndrome or patient has suspected Gilbert's Syndrome, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)

Exclusion Criteria:

1. Radiographic or cytologic evidence of leptomeningeal or multifocal disease at any time prior to study entry.
2. Prior conventional antitumor therapy, other than steroids, RT or TMZ therapy given for glioblastoma.
3. Pregnant or need to breast feed during the study period.
4. Not adhering to pregnancy prevention recommendations.
5. Active infection requiring intravenous antibiotics or an unexplained febrile (> 101.5 F) illness.
6. Immunosuppressive disease or human immunodeficiency virus infection.
7. Patients with unstable or severe intercurrent medical conditions such as severe heart or lung disease.
8. Allergic or unable to tolerate TMZ for any reason. Any patient that successfully completed at least 5 weeks of Temodar during standard of care XRT/TMZ and whose blood counts meet the eligibility requirements (inclusion #7) within 4 weeks post XRT/TMZ is eligible.
9. Patients with previous inguinal lymph node dissection, radiosurgery, brachytherapy, or radiolabeled monoclonal antibodies.
10. Prior allogeneic solid organ transplant.
11. Currently receiving or ever received immunosuppressive therapy for an autoimmune disorder or an organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ashley, MBBS, FRACP, PhD, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PEP-CMV vaccine originally was comprised of Component A (a pp65 synthetic long peptide [SLP]) and Component B (a neutralizing antibody epitope from human CMV glycoprotein B [gB] conjugated to KLH). Component B was removed due to insufficient manufacturing of Component B followed by hypersensitivity reactions in a subset of patients.
Period: Overall Study
Arm/Group | 5-day TMZ: Components A and B | 21-day TMZ: Components A and B | 5-day TMZ: Safety Cohort | 5-day TMZ: Component A Alone | 21-day TMZ: Component A Alone
Started | 4 | 1 | 6 | 8 | 8
Completed | 4 | 1 | 6 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-day TMZ: Components A and B | 21-day TMZ: Components A and B | 5-day TMZ: Safety Cohort | 5-day TMZ: Component A Alone | 21-day TMZ: Component A Alone | Total
Number analyzed (Participants) | 4 | 1 | 6 | 8 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.75 (8.14) | 40 (NA) — n=1 | 57.33 (9.97) | 57.63 (11.04) | 50.25 (8.84) | 55.19 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 2 | 4 | 11
  Male | 1 | 1 | 4 | 6 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 4 | 1 | 4 | 7 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 0 | 4 | 7 | 7 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-related Adverse Events
Description: To assess the safety of PEP-CMV vaccination in combination with adjuvant TMZ, the percentage of patients with unacceptable toxicity will be estimated within each arm. All patients who received any PEP-CMV vaccine will be included in these analyses.
Time Frame: 2 weeks after the 3rd vaccine, which is approximately 12 weeks after consent
Measure: Number; unit: percentage of participants
Arm/Group | 5-day TMZ: Components A and B | 21-day TMZ: Components A and B | 5-day TMZ: Safety Cohort | 5-day TMZ: Component A Alone | 21-day TMZ: Component A Alone
Number analyzed (Participants) | 4 | 1 | 6 | 8 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Immunologic Response as Measured by Peak Number of T Cells That Secrete IFNγ by ELISPOT in Response to Component A of PEP-CMV
Description: The primary analysis will focus on patients who have follow-up immunologic monitoring after the 3rd vaccination with component A alone and before initiation of the second TMZ/vaccine cycle. Such a patient is considered "evaluable" for the immunologic response primary analyses.
  The Wilcoxon rank sum test will compare treatment groups with regard to the median peak number of T cells that secrete IFNγ by ELISPOT in response to component A of PEP-CMV. Analyses will include only those patients who have an assessment of immune response after receiving 3 vaccinations.
Time Frame: Through study completion, an average of 1.5 years
Population: Participants who received Component A alone as well as an assessment of immune response after receiving 3 vaccinations. Data not collected on Components A and B cohorts or the Safety Cohort.
Measure: Median (Full Range); unit: T cells
Groups:
- 5-day TMZ: Components A and B: All patients receive Tetanus-Diphtheria booster vaccine at time of enrollment. Cycles of standard TMZ (150-200 mg/m^2/day on days 1-5 of each 28 day cycle) with PEP-CMV vaccination on Day 23 (-1 day, + 2 days) of each TMZ cycle and tetanus pre-conditioning the day before the first vaccine.
  5-day TMZ: Chemotherapy agent FDA approved to treat newly-diagnosed glioblastoma given as cycles of 150-200 mg/m^2/day on days 1-5 of each 28 day cycle PEP-CMV: Component A: 500 µg of PEP-CMV Component A (a synthetic long peptide) mixed with Montanide ISA-51 intradermally administered Tetanus-Diphtheria booster: At time of enrollment, after signing consent and undergoing immune monitoring blood work, patients will receive Tetanus-diphtheria booster vaccination with 0.5 mL of Td (tetanus, diphtheria toxoid, absorbed) Tetanus Pre-Conditioning: All patients will receive a tetanus pre-conditioning injection in the right groin intradermally on day 22 (±1 day) of the first post-radiation cycle of TMZ PEP-CMV: Component B: 500 µg of PEP-CMV Component B (a neutralizing antibody epitope from human CMV glycoprotein B conjugated to Keyhole Limpet Hemocyanin) mixed in 150 µg of GM-CSF intradermally administered
- 21-day TMZ: Components A and B: All patients receive Tetanus-Diphtheria booster vaccine at time of enrollment. Cycles of dose-intensified TMZ (75-100 mg/m^2/day on days 1-21 of each 28 day cycle) with PEP-CMV vaccination on day 23 (-1 day, + 2 days) of each TMZ cycle and tetanus pre-conditioning the day before the first vaccine.
  21-day TMZ: Chemotherapy agent FDA approved to treat newly-diagnosed glioblastoma given as cycles of dose-intensified TMZ (75-100 mg/m2/day on days 1-21 of each 28 day cycle) PEP-CMV: Component A: 500 µg of PEP-CMV Component A (a synthetic long peptide) mixed with Montanide ISA-51 intradermally administered Tetanus-Diphtheria booster: At time of enrollment, after signing consent and undergoing immune monitoring blood work, patients will receive Tetanus-diphtheria booster vaccination with 0.5 mL of Td (tetanus, diphtheria toxoid, absorbed) Tetanus Pre-Conditioning: All patients will receive a tetanus pre-conditioning injection in the right groin intradermally on day 22 (±1 day) of the first post-radiation cycle of TMZ PEP-CMV: Component B: 500 µg of PEP-CMV Component B (a neutralizing antibody epitope from human CMV glycoprotein B conjugated to Keyhole Limpet Hemocyanin) mixed in 150 µg of GM-CSF intradermally administered
- 5-day TMZ: Safety Cohort: All patients receive Tetanus-Diphtheria booster vaccine at time of enrollment. Cycles of standard TMZ (150-200 mg/m^2/day on days 1-5 of each 28 day cycle) with PEP-CMV vaccination on Day 23 (-1 day, + 2 days) of each TMZ cycle and tetanus pre-conditioning the day before the first vaccine. Vaccine components A and B were administered separately, with a delay between them, to determine if it was an individual component or a combination of the components that resulted in adverse reactions.
  5-day TMZ: Chemotherapy agent FDA approved to treat newly-diagnosed glioblastoma given as cycles of 150-200 mg/m^2/day on days 1-5 of each 28 day cycle PEP-CMV: Component A: 500 µg of PEP-CMV Component A (a synthetic long peptide) mixed with Montanide ISA-51 intradermally administered Tetanus-Diphtheria booster: At time of enrollment, after signing consent and undergoing immune monitoring blood work, patients will receive Tetanus-diphtheria booster vaccination with 0.5 mL of Td (tetanus, diphtheria toxoid, absorbed) Tetanus Pre-Conditioning: All patients will receive a tetanus pre-conditioning injection in the right groin intradermally on day 22 (±1 day) of the first post-radiation cycle of TMZ PEP-CMV: Component B: 500 µg of PEP-CMV Component B (a neutralizing antibody epitope from human CMV glycoprotein B conjugated to Keyhole Limpet Hemocyanin) mixed in 150 µg of GM-CSF intradermally administered
Arm/Group | 5-day TMZ: Components A and B | 21-day TMZ: Components A and B | 5-day TMZ: Safety Cohort | 5-day TMZ: Component A Alone | 21-day TMZ: Component A Alone
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 4
T cells |  |  |  | 57.5 [13.5 to 241.5] | 71.25 [28 to 146]

3. Secondary Outcome: Antigen Loss
Description: To determine if tumors are CMV antigen negative by immunohistochemical analysis for the presence of the antigen pp65 at the time of disease progression/recurrence
Time Frame: Through study completion, an average of 1.5 years
Population: No data collected with respect to this outcome. Tumor was not collected at the time of disease progression/recurrence.
Arm/Group | 5-day TMZ: Component A Alone | 21-day TMZ: Component A Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 Months
Arm/Group | 5-day TMZ: Components A and B | 21-day TMZ: Components A and B | 5-day TMZ: Safety Cohort | 5-day TMZ: Component A Alone | 21-day TMZ: Component A Alone
All-Cause Mortality (participants affected / at risk) | 4/4 | 1/1 | 6/6 | 8/8 | 8/8
Serious Adverse Events (participants affected / at risk) | 4/4 | 1/1 | 2/6 | 6/8 | 4/8
Other Adverse Events (participants affected / at risk) | 4/4 | 1/1 | 6/6 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-day TMZ: Components A and B (N=4) | 21-day TMZ: Components A and B (N=1) | 5-day TMZ: Safety Cohort (N=6) | 5-day TMZ: Component A Alone (N=8) | 21-day TMZ: Component A Alone (N=8)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 3 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 2 | 0
Fever (General disorders) | 1 | 0 | 0 | 1 | 0
Flu like symptoms (General disorders) | 1 | 0 | 0 | 4 | 4
Cytokine release syndrome (Immune system disorders) | 2 | 1 | 0 | 0 | 0
Infections and infestations - Other, Specify: PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Investigations - Other, Specify: LACTIC ACIDOSIS (Investigations) | 0 | 0 | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 | 2 | 0
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 3 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-day TMZ: Components A and B (N=4) | 21-day TMZ: Components A and B (N=1) | 5-day TMZ: Safety Cohort (N=6) | 5-day TMZ: Component A Alone (N=8) | 21-day TMZ: Component A Alone (N=8)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 5 | 6 | 5
Blood and lymphatic system disorders - Other, Specify: CUT FACE SHAVING; BLED FOR 2+ HOURS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0 | 3 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ear and labyrinth disorders - Other, Specify: "CLOGGED FEELING" (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 2
Eye disorders - Other, Specify: LEFT EYE WEEPY, RED, SWOLLEN, BLOOD SHOT (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, Specify: RED, ITCHY EYES (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, Specify: REDNESS (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, Specify: REQUIRES BRIGHTER LIGHTS WHEN INSIDE IN ORDER TO SEE (Eye disorders) | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, Specify: CRAMPING (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 5 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 1
Chills (General disorders) | 1 | 0 | 4 | 3 | 0
Edema limbs (General disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 4 | 3 | 1
Fever (General disorders) | 0 | 0 | 2 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 2 | 2
Gait disturbance (General disorders) | 0 | 0 | 0 | 3 | 1
General disorders and administration site conditions - Other, Specify: NIGHT SWEATS (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 2 | 1 | 4 | 7 | 6
Pain (General disorders) | 0 | 0 | 2 | 2 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 2 | 0 | 5 | 6 | 4
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other, Specify: SHINGLES (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 2 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 3 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 2 | 1 | 1
Lymphocyte count decreased (Investigations) | 2 | 0 | 3 | 7 | 5
Neutrophil count decreased (Investigations) | 1 | 0 | 4 | 3 | 2
Platelet count decreased (Investigations) | 1 | 0 | 1 | 5 | 4
White blood cell decreased (Investigations) | 1 | 0 | 3 | 3 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 8 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 4 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 5 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 4 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Metabolism and nutrition disorders - Other, Specify: NIGHT SWEATS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified - Other, Specify: SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 2 | 2 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 5 | 2 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 3 | 1 | 0
Nervous system disorders - Other, Specify: A LITTLE WOBBLY, OFF BALANCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nervous system disorders - Other, Specify: HEMIANOPSIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nervous system disorders - Other, Specify: QUADRANTANOPSIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 1 | 4 | 1
Seizure (Nervous system disorders) | 0 | 0 | 2 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 4 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, Specify: "LUMP IN THROAT" (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, Specify: "STRANGE SENSATION ON THROAT" (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, Specify: DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Skin and subcutaneous tissue disorders - Other, Specify: DARK CRUSTY SPOTS POSS. ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 — Top of head
Skin and subcutaneous tissue disorders - Other, Specify: FEVER BLISTER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Specify: POISON IVY (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Specify: POSSIBLE PRECANCEROUS LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 4 | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 1
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 5 | 5 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol Document with SAP (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT02864368/Prot_SAP_000.pdf